CLINICAL TRIAL: NCT05710614
Title: Mixed Plant- vs. Animal-based Supplementary Protein to Support Muscle Adaptations to Resistance Exercise: a Randomized Clinical Trial
Brief Title: Distinct Sources of Supplementary Protein in the Resistance Exercise Training-induced Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: NotCo Brasil Distribuicao e Comercio de Produtos Alimenticios LTDA (Unknown)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, Doctor of Philosophy, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66029522.3.0000.0068
Record Dates: First submitted 2023-01-20; First posted 2023-02-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dietary Supplements; Muscle Strength; Muscle, Skeletal; Resistance Training; Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Plant Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- animal protein (Active Comparator): Whey protein will be used as the active comparator for animal protein arm
  Interventions: Dietary Supplement: Animal protein
- plant protein (Experimental): A combination of pea and soy protein will be used as the experimental arm
  Interventions: Dietary Supplement: Plant Protein

INTERVENTIONS:
Dietary Supplement: Animal protein — Patients allocated to this arm will be submitted a supervised resistance training program in combination with the intake of three 15-g daily doses (45g. d- 1 total) animal-based protein (i.e.; whey protein) in drink form as a supplementary source of protein in their main meals of the day.
  Arms: animal protein
Dietary Supplement: Plant Protein — Patients allocated to this arm will be submitted a supervised resistance training program in combination with the intake of three 15-g daily doses (45g. d- 1 total) mixed plant protein (i.e.; soy and pea) in drink form as a supplementary source of protein in their main meals of the day.
  Arms: plant protein

SUMMARY:
This is a randomized controlled trial aimed to investigate the effects of different supplementary protein sources on muscle adaptations to resistance exercise. Young, healthy, recreationally active participants consuming an omnivorous diet with protein intake within recommended dietary allowance (RDA) (i.e.; 0.8-1.0 g.kg-1. d-1) will be recruited to undergo a 12-wk supervised resistance training program in combination with the intake of three 15-g daily doses (45g. d-1 total) of either a mixed plant- (i.e.; soy and pea protein) or animal-based (i.e.; whey protein) protein in drink form as a supplementary source of protein to their main meals of the day (i.e.; breakfast, lunch, and dinner). Before (PRE) and after (POST) the 12-wk intervention, participants will be assessed for body composition by dual-energy X-ray absorptiometry (DXA), muscle cross-sectional area (ultrasound) and fiber cross-sectional area (muscle biopsy), and maximal isotonic strength (1RM). Training consists of a resistance training (RT) program individually supervised by a researcher blinded to treatment in a laboratorial setting. Assessments will also be conducted in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (according to the International Physical Activity Questionnaire (IPAQ)
* Absence of any chronic condition that could preclude participation in a RT program or physical testing
* Habitual protein consumption within RDA ≥ 0.8 ≤1.0 g.kg-1. d-1

Exclusion Criteria:

* Prior history of anabolic steroids use, current or previous (≤ 3 m)
* Use of ergogenic or protein-based supplements, current or previous (< 1 y)
* Engagement in energy-restricted diets

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
vastus lateralis muscle cross sectional area | Ultrasound images will be obtained both at baseline (before the comencement of the study) and immediately after the 12-week intervention period
  the investigators used ultrasound measures of the vastus lateralis cross sectional area as the primary outcome

SECONDARY OUTCOMES:
lean mass | DXA scans will be taken both at baseline (before the comencement of the study) and immediately after the 12-week intervention period
  total body and lower limb lean mass assessed by DXA
fiber cross sectional area | Fiber cross sectional areas will be measured both at baseline (before the comencement of the study) and immediately after the 12-week intervention period
  vastus lateralis fiber cross sectional area from muscle biopsy samples
maximal isotonic strength | 1-RM tests will be taken both at baseline (before the comencement of the study) and immediately after the 12-week intervention period
  lower-limb maximal isotonic strength will be assessed in the leg-press exercise by means of the one-repetition-maximum test (1-RM test)

CONTACTS AND LOCATIONS:
Overall Officials: Hamilton Roschel, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santini MH, Erwig Leitao A, Mazzolani BC, Smaira FI, de Souza MSC, Santamaria A, Gualano B, Roschel H. Similar effects between animal-based and plant-based protein blend as complementary dietary protein on muscle adaptations to resistance training: findings from a randomized clinical trial. J Int Soc Sports Nutr. 2025 Dec;22(1):2568047. doi: 10.1080/15502783.2025.2568047. Epub 2025 Oct 8. PMID 41059835